CLINICAL TRIAL: NCT02532062
Title: Efficacy of Vitamin D Supplementation in Vitamin D-deficient Subjects at Risk of Lung Cancer (The Pittsburgh Vitamin D Study)
Brief Title: The Pittsburgh Vitamin D Study: Vitamin D Supplementation in Vitamin D-deficient Subjects at Risk of Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lost funding, limited eligibility due to pre-existing vitamin D supplementation
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David O. Wilson, MD, MPH, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PRO15020031; P50CA090440 (NIH)
Record Dates: First submitted 2015-08-11; First posted 2015-08-25 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Deficiency of Vitamin D3; COPD
Keywords: lung cancer risk; cigarette smokers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplementation (Experimental): Participants who are assigned to the Supplementation arm will receive a vitamin D supplement containing 4,000 units of vitamin D3 (cholecalciferol; capsule form) plus an oral multivitamin containing 400 units of vitamin D3 daily for a period of one year.
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: multivitamin
- Placebo (Active Comparator): Participants who are assigned to the Placebo arm will receive a placebo supplement plus an oral multivitamin containing 400 units of vitamin D3 daily for a period of one year.
  Interventions: Dietary Supplement: multivitamin; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 4,000 IU, oral, once a day for one year
  Other Names: Vitamin D3
  Arms: Supplementation
Dietary Supplement: multivitamin — oral, once a day for one year
Dietary Supplement: Placebo — oral, once a day for one year
  Arms: Placebo

SUMMARY:
This study aims to establish the ability of 4,000 IU oral vitamin D3 per day (in combination with a daily multivitamin) to safely convert vitamin D3-deficient subjects at increased risk of lung cancer to a vitamin D3-sufficient state, and to explore effects of vitamin D3 supplementation in this population on markers of inflammation and lung cancer risk. Current and former smokers with chronic obstructive pulmonary disease (COPD) are at increased risk of developing lung cancer and represent the clinical population of interest for this study.

DETAILED DESCRIPTION:
Smoking avoidance or cessation are essential to the prevention of lung cancer. However, not all smokers are able to quit smoking and, importantly, former smokers remain at increased risk of lung cancer compared to never smokers. Despite smoking prevention/cessation programs and treatment advances, lung cancer is still the leading cause of cancer-related mortality in the United States with more than 158,000 individuals expected to die from this disease in 2015. Effective and safe prevention strategies are expected to be more successful in reducing lung cancer deaths than treatment of established disease.

NF-kappaB (NF-kB) pathway activation underlies smoking-related inflammation and lung carcinogenesis, and those agents which suppress NF-κB signaling may have the potential to prevent lung cancer. Recent preclinical data from our group and others indicate that the active metabolite of vitamin D3, 1,25-dihydroxyvitamin D3 [1,25(OH)2D3], has lung cancer chemopreventive activity. Because systemic 1,25(OH)2D3 administration is complicated by its hypercalcemia-inducing properties, the investigators propose to use oral supplementation with vitamin D3 (cholecalciferol) to safely achieve chemopreventive 1,25(OH)2D3 levels within the lung.

This randomized, placebo-controlled Phase IIb study aims to evaluate the ability of 4,000 IU oral vitamin D3/day (in combination with a daily multivitamin) to safely convert vitamin D3-deficient subjects at risk of lung cancer to a vitamin D3-sufficient state.

Study participants will be recruited from among Pittsburgh Lung Screening Study Extension (PLuSS-X) and PLuSS-XX participants not diagnosed with lung cancer, and from among the patient population seen by the PI of this protocol. The study consists of two stages, a screening and an intervention stage, with their own consent forms. In Stage 1 (the screening stage), the vitamin D3 status of subjects potentially eligible for participation in the intervention will be determined; in Stage 2 (the intervention stage), supplementation with oral vitamin D3 will be evaluated.

Participants who fulfill the eligibility criteria and provided signed consent for Stage 2 will be randomized in a 2:1 ratio to receive: (A) 4,000 IU vitamin D3 plus a multivitamin (containing 400 IU vitamin D3) daily for one year, or (B) a placebo vitamin D3 pill plus a multivitamin daily for one year. Both groups will contain equal numbers of current and ex-smokers; in total 120 subjects will be randomized. To evaluate whether supplementation safely corrects vitamin D3 deficiency in this population, blood samples will be obtained at baseline, 3, 6, and 12 months of intervention for evaluation of 25(OH)D3 and serum calcium. The collected blood will also be used to facilitate biomarker assessment. Pulmonary function tests (PFTs) will be obtained at baseline and repeated after 12 months to determine whether supplementation has an effect on lung function. Sputum and nasal epithelium will be collected at baseline, 6 months and 12 months to facilitate biomarker assessment.

- Study Objectives Primary Objective: To establish the 12-month conversion rate (i.e., proportion of subjects whose baseline vitamin D3 deficiency is corrected after 12 months of supplementation).

Secondary Objectives: To determine the 3-month and 6-month conversion rates and examine the effect of vitamin D3 supplementation in current and former smokers. Additionally, to examine the effects of vitamin D3 supplementation on biomarkers of lung cancer risk, inflammation, and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years old.
2. Current or ex-smoker with at least 10 pack-year history
3. COPD, GOLD II or greater (defined as FEV1/FVC <70% and FEV1 % predicted <80%)
4. 25(OH)D3 level ≤25 ng/mL
5. Willingness to comply with study guidelines.
6. Willingness to avoid alternative/additional vitamin D3 supplementation for the duration of the trial
7. Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

1. Personal history of lung cancer or head and neck cancer
2. History of malabsorption syndrome (e.g., pancreatic insufficiency, celiac disease, or tropical sprue).
3. History of known thyroid disease
4. History of known sarcoid disease
5. History of known abnormalities in calcium metabolism
6. Hypercalcemia (serum calcium in excess of laboratory ULN)
7. Self-reported consumption of more than 4 alcoholic drinks per day
8. Use of anti-seizure medications phenobarbital or phenytoin, which can disrupt vitamin D metabolism
9. History of known renal dysfunction
10. History of known nephrolithiasis (kidney stones)
11. Current participation in another cancer chemoprevention study
12. Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to receive study drug.
13. Inability to swallow pills.
14. Vitamin D supplementation > 2,000 IU/day of vitamin D within 30 days prior to enrollment.
15. Being pregnant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
The 12-month conversion rate | 12 months
  The proportion of subjects whose baseline vitamin D3 deficiency is corrected after 12 months of supplementation (i.e., the 12-month conversion rate).

SECONDARY OUTCOMES:
The 3-month conversion rate | 3 months
The 6-month conversion rate | 6 months
Pulmonary function as measured by spirometry | 12 months
  Effect of vitamin D supplementation on lung function as measured by spirometry will be evaluated.
Promoter methylation status in sputum and nasal swab samples | 12 months
  Effect of supplementation on promoter methylation status of genes previously reported associated with lung cancer risk (e.g., RAMP2, p16, MGMT) in sputum and nasal swab samples will be explored.
Protein expression in sputum and nasal swab samples | 12 months
  Effect of supplementation on the expression of proteins, including inflammation and vitamin D metabolism-related proteins, in sputum and nasal swab samples will be explored.
Concentration of inflammatory markers in blood | 12 months
  Blood samples will be analyzed for inflammatory markers such as IL6 and CRP and the effect of supplementation on the examined cytokines will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: David Wilson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided